CLINICAL TRIAL: NCT03546465
Title: A Phase 1 Bridging Study to Investigate and Compare the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Four Single Ascending Doses of Ropeginterferon Alfa-2b (P1101) in Healthy Japanese and Healthy Caucasian Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics & Pharmacodynamics Study of Ropeginterferon Alfa-2b in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia Japan K.K. (Industry)
Collaborators: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A17-102
Record Dates: First submitted 2018-05-06; First posted 2018-06-06 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohorts 1C (Caucasian subjects) (Experimental): ropeginterferon alfa-2b: single dose of 100 μg
  Interventions: Drug: ropeginterferon alfa-2b
- Cohorts 1J (Japanese subjects) (Experimental): ropeginterferon alfa-2b: single dose of 100 μg
  Interventions: Drug: ropeginterferon alfa-2b
- Cohorts 2C (Caucasian subjects) (Experimental): ropeginterferon alfa-2b: single dose of 200 μg
  Interventions: Drug: ropeginterferon alfa-2b
- Cohorts 2J (Japanese subjects) (Experimental): ropeginterferon alfa-2b: single dose of 200 μg
  Interventions: Drug: ropeginterferon alfa-2b
- Cohorts 3C (Caucasian subjects) (Experimental): ropeginterferon alfa-2b: single dose of 300 μg
  Interventions: Drug: ropeginterferon alfa-2b
- Cohorts 3J (Japanese subjects) (Experimental): ropeginterferon alfa-2b: single dose of 300 μg
  Interventions: Drug: ropeginterferon alfa-2b
- Cohorts 4C (Caucasian subjects) (Experimental): ropeginterferon alfa-2b: single dose of 450 μg
  Interventions: Drug: ropeginterferon alfa-2b
- Cohorts 4J (Japanese subjects) (Experimental): ropeginterferon alfa-2b: single dose of 450 μg
  Interventions: Drug: ropeginterferon alfa-2b

INTERVENTIONS:
Drug: ropeginterferon alfa-2b — 6 subjects in each cohort will receive a single dose by subcutaneous injection
  Other Names: P1101

SUMMARY:
This is a Phase 1 single center, parallel group study to assess and compare the safety, tolerability, PK and PD of 4 single ascending doses of P1101 (100, 200, 300, and 450 μg) following subcutaneous administration in healthy Japanese and Caucasian subjects.

DETAILED DESCRIPTION:
Twenty-four healthy eligible Japanese male subjects and 24 healthy eligible Caucasian male subjects, each divided into 4 cohorts of 6 subjects, will participate in this study. No subject will participate in more than 1 cohort and all subjects will receive a single dose of P1101. Caucasian subjects will be body weight- and height-matched to Japanese subjects.

Dosing will be initiated with the lowest dose of 100 μg in both Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all of the following criteria apply:

* Adult Japanese and Caucasian males aged 21 to 50 years inclusive and body mass index (BMI) between 19 and 30 kg/m2.
* Japanese subjects must be first generation (born in Japan) with parents and grandparents born in Japan, lived for < 10 years outside of Japan, and have no significant change in life style since leaving Japan.
* Caucasian subjects must have both parents of Caucasian descent; Caucasian subjects are defined as descendants of the original peoples of Europe.
* Individual Caucasian subjects should be selected to match body weight (± 20%) and height (± 15%) of corresponding Japanese subjects.
* Subjects must be willing to use effective methods of contraception during the entire study period and for 12 weeks after dosing on Day 1.
* Subjects who are healthy as determined by pre-study medical history, physical examination, and 12-lead ECG.
* Subjects whose clinical laboratory test results are within the reference ranges for hematological parameters and liver function tests at Screening and Day -1. For results outside the reference range at Screening and considered not clinically significant by the Investigator a repeat test is allowed once during the Screening period. Note: subjects with an absolute neutrophil count below 2.0 × 109/L will be excluded. All other clinical laboratory test results must be within the reference range or judged not to be clinically significant and acceptable to the Investigator.
* Subjects whose thyroid function tests are within the study reference range.
* Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus antibody (HCVAb) and human immunodeficiency virus (HIV) I and II tests at Screening.
* Subjects who are negative for drugs of abuse and alcohol tests at Screening. Alcohol will be measured using breathalyzer test. If the tests are negative at Screening, and if they meet other eligibility criteria, the subject may be included. A repeat test for suspected false positive at Screening (with documented rationale) may be performed at the discretion of the Investigator. However, if the tests are subsequently positive on Admission, the subject should be withdrawn from the study. Repeat tests are not allowed at Admission.
* Subjects who are non-smokers for at least 6 months preceding Screening.
* Subjects who are able and willing to give a valid written informed consent.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

* Subjects who do not conform to the above inclusion criteria.
* Female subjects.
* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, coagulation, endocrine, lymphatic, neurological, cardiovascular, psychiatric, ophthalmological, musculoskeletal, genitourinary, immunological, autoimmune, dermatological, and connective tissue diseases or disorders.
* Subjects who have a first degree relative with autoimmune disease (e.g. thyroiditis, lupus, rheumatoid arthritis, etc.) or other clinically relevant medical history which in the opinion of the Investigator poses a risk to the subject.
* Subjects with a history of latent or active tuberculosis or exposure to endemic areas.
* Subjects with a positive result in the QuantiFERON-TB Gold test and/or clinically significant abnormality on chest X-ray.
* Subjects who have a clinically relevant surgical history and history of any prior malignancy.
* Subjects who, in the opinion of the Investigator, have clinically relevant medical history in their immediate family (first degree relative).
* Subjects with current symptoms of eczema or hay fever, or subjects with a history of hay fever requiring medication when their hay fever season starts within the expected duration of the study.
* Subjects who have a history of severe allergy and severe drug reaction (e.g., anaphylaxis, or other drug reaction requiring hospitalization to beta lactam antibiotics OR any other relevant drug hypersensitivity).
* Subjects who have a history of alcoholism.
* Subjects who consume more than the recommended number of 14 units of alcohol per week. (1 unit = 1 glass of wine [125 mL] = 1 measure of spirits = ½ pint of beer).
* Subjects who have a history of drug abuse.
* Subjects who have abnormal vital signs, after 10 minutes supine rest (measurements may be repeated after 15 minutes at the discretion of the Investigator where they suspect that the initial values are not representative of the usual values due to some factors e.g., anxiety), defined as any of the following at Screening:

  1. Systolic blood pressure < 90 mmHg or ≥ 140 mmHg;
  2. Diastolic blood pressure < 50 mmHg or ≥ 90 mmHg;
  3. Pulse rate < 40 or > 100 beats per minute.
* Subjects who have any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes.
* Subjects who have a prolonged QTcF > 450 ms or family history of long QT syndrome.
* Subjects who have a significant infection such as a respiratory infection or known inflammatory process at Screening or Admission.
* Subjects who have a clinically significant history or evidence of any active or suspected bacterial, viral, fungal or parasitic infection within the 30 days prior to Admission (e.g., common cold, viral syndrome, flu-like symptoms, etc).
* Subjects who have acute gastrointestinal symptoms at Screening or Admission (e.g., nausea, vomiting, diarrhea, and heartburn).
* Subjects who have used 1 or more prescription drugs within 28 days prior to Day 1.
* Subjects who have used non-prescription drugs or other products (supplements, herbal preparations, etc) with enzyme inducing properties such as St John's Wort within 28 days prior to the first administration of investigational product.
* Subjects who have used other non-prescription drugs excluding routine vitamins but including megadose (intake of 20 to 600 times the recommended daily dose) vitamin therapy within 7 days of first administration of investigational product, unless agreed as not clinically relevant by the Principal Investigator and Sponsor.
* Subjects who have received any live vaccine in the 6 months prior to Screening.
* Subjects who have previously been exposed to interferon or peginterferon.
* Subjects who have received the last dose of investigational product within the last 3 months or within 5 times the half-life, whichever is longer and those who are on extended follow-up.
* Subjects who are vegans or have medical dietary restrictions.
* Subjects who have consumed grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of investigational product.
* Subjects who have donated blood/plasma within 3 months of Screening or who have had any blood loss > 500 mL during the 3 months prior to Screening.
* Subjects who are staff members at the investigational site.
* Subjects who are Contract Research Organization staff members, Sponsor employees, and affiliates.
* Subjects who cannot understand or communicate reliably with the Investigator.
* Subjects who are unlikely to co-operate with the requirements of the study.
* Subjects who have been shown to have a suicidal tendency following completion of the C-SSRS.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Adverse events after single dose | Through study Day 35
  Frequency and severity of all adverse events among subjects, including frequency and severity of drug-related adverse events.
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration [AUC(0-last)]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Area under the plasma concentration-time curve from time zero extrapolated to infinity [AUC(0-inf)]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Observed maximum plasma concentration [Cmax]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Time to reach Cmax [tmax]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  apparent terminal rate constant
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Apparent terminal half-life [t½]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Apparent systemic clearance [CL/F]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  apparent volume of distribution during the terminal phase [Vz/F]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  dose normalized AUC(0-last) [AUC(0-last)/Dose]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  dose normalized AUC(0-inf) [AUC(0-inf)/Dose]
Pharmacokinetics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Dose normalized Cmax [Cmax/Dose]

SECONDARY OUTCOMES:
Pharmacodynamics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Beta-2 microglobulin: maximum serum biomarker response [Emax]
Pharmacodynamics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Beta-2 microglobulin: time to Emax [TEmax]
Pharmacodynamics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Beta-2 microglobulin: area under the serum biomarker effect-time curve [AUEC(0-t)]
Pharmacodynamics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Neopterin: maximum serum biomarker response [Emax]
Pharmacodynamics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Neopterin: time to Emax [TEmax]
Pharmacodynamics of ropeginterferon alfa-2b after single dose | Through study Day 35
  Neopterin: area under the serum biomarker effect-time curve [AUEC(0-t)]

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Qin A, Shimoda K, Suo S, Fu R, Kirito K, Wu D, Liao J, Chen H, Wu L, Su X, Gao Y, Sato T, Li Y, Zhang J, Shen W, Wang W, Zhang L, Jin J, Komatsu N. Population Pharmacokinetics-Pharmacodynamics and Exposure-Response of Ropeginterferon Alfa-2b in Chinese and Japanese Patients With Polycythemia Vera. Pharmacol Res Perspect. 2025 Jun;13(3):e70109. doi: 10.1002/prp2.70109. PMID 40313042
- [Derived] Miyachi N, Zagrijtschuk O, Kang L, Yonezu K, Qin A. Pharmacokinetics and Pharmacodynamics of Ropeginterferon Alfa-2b in Healthy Japanese and Caucasian Subjects After Single Subcutaneous Administration. Clin Drug Investig. 2021 Apr;41(4):391-404. doi: 10.1007/s40261-021-01026-5. Epub 2021 Mar 16. PMID 33725322